CLINICAL TRIAL: NCT05414331
Title: WithDRawal Impact Of Postoperative Beta-Blocker
Acronym: DROP-BB
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated as both investigators left the institution.
Sponsor: Yale University (Other)
Collaborators: Glenn Memorial Fund (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2000032771
Record Dates: First submitted 2022-06-07; First posted 2022-06-10 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Coronary Artery Bypass
Keywords: beta-blocker

STUDY DESIGN:
Intervention Model Description: Aim 1: The investigators will enroll patients with preserved EF (EF ≥50%) who underwent isolated elective or non-elective CABG at Yale New Haven Hospital (YNHH). Blocked randomization will be applied to ensure an equal sample size. Patients will be randomized to 1) continuation of the current BB regimen and 2) discontinuation of all BB, and medication changes will be made at the 1-month clinic visit. A cardiopulmonary exercise test (CPET) will be performed 1 month after the randomization (2 months after CABG).
  Aim 2: Patients will be randomized at a 1-month postoperative visit, and the outcome will be adjudicated at 12 months since CABG.
  The safety endpoint is all-cause death, myocardial infarction, stroke, or repeat revascularization at 12 months. The investigators will measure patient-reported outcome on 1) 10-item activity level (VSAQ), 2) Fatigue Assessment Scale. 3) 15-item Vertigo Symptom Scale at the time of enrollment and 3 months.
Masking Description: Blinding will be only on the investigator interpreting CPET and adjudicating major cardiac and cerebrovascular events
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continuation of beta-blocker regimen (No Intervention): Participants will continue with current standard of care on current beta-blocker regimen
- Withdrawing of beta-blockers (Experimental): Discontinuation of all BB, and medication changes will be made at the 1-month clinic visit. A cardiopulmonary exercise test (CPET) will be performed 1 month after the randomization (2 months after CABG).
  Interventions: Other: Discontinuing all beta-blocker

INTERVENTIONS:
Other: Discontinuing all beta-blocker — All beta-blockers will be stopped 2 months after CABG
  Arms: Withdrawing of beta-blockers

SUMMARY:
The investigators will evaluate the impact of withdrawing beta-blocker medication after coronary artery bypass surgery with this randomized controlled trial.

DETAILED DESCRIPTION:
Aim 1: The primary aim is to evaluate the impact of withdrawing BB on exercise capacity (peak oxygen consumption, VO2 max) in patients who underwent CABG. The investigators hypothesize that withdrawing BB 1 month after CABG will improve exercise capacity 2 months after CABG.

Aim 2: The secondary objectives are to evaluate the impact of withdrawing BB on a MACCE (major adverse cardiac and cerebrovascular event) and fatigue-related symptoms in patients who underwent CABG. The investigators hypothesize that withdrawing BB after CABG for 1 year will be non-inferior to continuing BB in terms of MACCE incidence.

ELIGIBILITY:
Inclusion Criteria:

* Participants who underwent coronary artery bypass graft(CABG) surgery at Yale New Haven Hospital who presented to 1-month postoperative visit
* ejection fraction >50%, and in sinus rhythm at the time of hospital discharge or enrollment.

Exclusion Criteria:

* those who underwent combined valve + CABG surgery or aorta + CABG surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Peak oxygen consumption (VO2 max) to measure cardiorespiratory fitness | 1 month
  Peak oxygen measured in ml/kg/min consumption will be measured on CPET 1 month after randomization and be compared controls. This is an important measure of exercise capacity, which has been shown to decrease in other population when on beta-blocker. The higher the measure, the better with measures greater than 12.3 ml/kg/min as positive.

SECONDARY OUTCOMES:
Adherence to medication and adjudication of endpoint | 3 months
  Phone follow-ups at 3 months after CABG to ensure medication adherence and to adjudicate whether the endpoint had occurred
Adherence to medication and adjudication of endpoint | 6 months
  Phone follow-ups at 6 months after CABG to ensure medication adherence and to adjudicate whether the endpoint had occurred
Adherence to medication and adjudication of endpoint | 12 months
  Phone follow-ups at 12 months after CABG to ensure medication adherence and to adjudicate whether the endpoint had occurred
Change in activity level measured using the Veterans Specific Activity Questionnaire(VSAQ) | baseline and 3 months
  VSAQ, a 10-item self reported questionnaire will be used to assess activity levels. Participants choose which item best describes their condition best. Items range from 1(low activity) to 13(higher activity). The higher the score, the more active.
Change in fatigue measured using the Fatigue Assessment Scale (FAS) | baseline and 3 months
  The FAS is a self reported 10-item general fatigue questionnaire to assess fatigue. Five questions reflect physical fatigue and 5 questions (questions 3 and 6-9) mental fatigue. The total score ranges from 10 to 50. A total FAS score < 22 indicates no fatigue, a score ≥ 22 indicates fatigue.
Change in vertigo symptoms measured using the Vertigo Symptom Scale-short form | baseline and 3 months
  The 15-item short form self report Vertigo Symptom Scale will be used to assess symptoms: 8 items relating to vertigo-balance, and 7 items relating to autonomic-anxiety symptoms. Each item is scored on a 5-point scale (range 0-4) and the total scale score ranges 0-60 with higher scores indicating more severe problems. Severe dizziness indicated by a score of ≥ 12 points .

CONTACTS AND LOCATIONS:
Overall Officials: Arnar Geirsson, MD, Principal Investigator — Yale University; Makoto Mori, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No